CLINICAL TRIAL: NCT05760079
Title: A Pilot Study of Lactoferrin Among Patients Reporting Taste or Smell Abnormalities After COVID-19
Brief Title: Lactoferrin for COVID-19-Induced Taste or Smell Abnormality
Acronym: TSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult to coordinate between all of the different support systems needed across various departments
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00074029
Record Dates: First submitted 2023-03-03; First posted 2023-03-08 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-06

CONDITIONS: Covid19; Taste Disorder, Secondary; Taste Disorders; Dysgeusia; Smell Disorder; Ageusia; Anosmia
Keywords: Lactoferrin; Taste disorder; Smell disorder; COVID-19
MeSH Terms: conditions — COVID-19; Taste Disorders; Dysgeusia; Olfaction Disorders; Ageusia; Anosmia | interventions — Lactoferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lactoferrin Supplementation (Experimental): 750mg lactoferrin (three 250mg tablets) per day for 30 days
  Interventions: Dietary Supplement: Lactoferrin

INTERVENTIONS:
Dietary Supplement: Lactoferrin — 750mg of Jarrow formulas taken three times daily for 30 days
  Other Names: Jarrow Formulas Apolactoferrin

SUMMARY:
Common side effects of corona virus disease 2019 (COVID-19) include disruptions in taste and smell function, which may persist for prolonged periods of time following recovery and resolution of COVID-19 infection. These disruptions not only reduce the hedonic pleasure derived from eating, but may also be detrimental to quality of life and could pose additional health risks (malnutrition) among patients with chronic illness or those enduring long-term complications from their previous COVID-19 infection.

Previous studies conducted among patients with cancer experiencing taste and smell abnormalities have indicated improvement in taste and smell function following daily lactoferrin supplementation. Lactoferrin is a natural transferrin protein that scavenges and chelates iron byproducts produced as a function of lipid oxidation in the oral cavity following inflammation, infection, or toxicity of chemosensory tissues.

The purpose of this pilot investigation is to assess the feasibility and preliminary effectiveness of lactoferrin supplementation (750mg per day for 30 days) for the treatment of taste and smell disturbances following COVID-19 infection.

Approximately 40 patients who experienced disruptions in taste and smell following infection with COVID-19 will be recruited. Participants will complete baseline assessments (questionnaires, blood draw) and will be given 90 lactoferrin tablets (provided by Jarrow Formulas) in order to take 3 tablets per day for 30 days.

DETAILED DESCRIPTION:
Common side effects of corona virus disease 2019 (COVID-19) include disruptions in taste and smell function, which may persist for prolonged periods of time following recovery and resolution of COVID-19 infection. These disruptions not only reduce the hedonic pleasure derived from eating, but may also be detrimental to quality of life and could pose additional health risks (malnutrition) among patients with chronic illness or those enduring long-term complications from their previous COVID-19 infection.

Previous studies conducted among patients with cancer experiencing taste and smell abnormalities have indicated improvement in taste and smell function following daily lactoferrin supplementation. Lactoferrin is a natural transferrin protein that scavenges and chelates iron byproducts produced as a function of lipid oxidation in the oral cavity following inflammation, infection, or toxicity of chemosensory tissues.

The purpose of this pilot investigation is to assess the feasibility and preliminary effectiveness of lactoferrin supplementation (750mg per day for 30 days) for the treatment of taste and smell disturbances following COVID-19 infection. Primary outcomes will be subjective change in taste and smell abnormalities obtained via the Taste and Smell Questionnaire (TSQ).

Approximately 40 patients who experienced disruptions in taste and smell following infection with COVID-19 will be recruited. Participants will complete baseline assessments. Participants will be given 90 lactoferrin tablets (provided by Jarrow Formulas) in order to take 3 tablets per day for 30 days. Primary outcomes will be assessed immediately following the 30 day supplementation period. After 30 additional days without lactoferrin supplements (a washout period), participants will complete follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* adult aged 18 or older; diagnosis of COVID-19 in the past 6 months; self-reported disruption in taste and smell beginning after infection with COVID-19

Exclusion Criteria:

* remains infectious from Covid-19; pregnant or lactating; taste or smell disruption existed prior to covid-19 infection; has cancer or is receiving cancer therapy; milk and/or iron allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in Taste disruption Scores | Baseline to day 60
  Ageusia or dysgeusia determined by subjective Smell and Taste Questionnaire (TSQ). As part of the questionnaire, participants will be asked to rate their individual taste and smell abnormalities as "insignificant," "mild," "moderate," "severe," or "incapacitating." The tool yields a taste complaint score (0-10) on the basis of subject responses to nine questions addressing changes to the sense of taste. One point is added for each reported taste complaint and two points for a rating of "severe" or "incapacitating" on the severity of the taste abnormality question.
Change in Smell disruption Scores | Baseline to day 60
  Anosmia or Dysnosmia determined by subjective Smell and Taste Questionnaire (TSQ). As part of the questionnaire, participants will be asked to rate their individual taste and smell abnormalities as "insignificant," "mild," "moderate," "severe," or "incapacitating." The tool yields a taste complaint score (0-6) on the basis of subject responses to five questions addressing changes to the sense smell. A smell complaint score (0-6) will be generated by adding one point for a positive response to each of five questions addressing self-perceived changes to the sense of smell. Two points will be assigned to a severity rating of "severe" or "incapacitating" for the severity of the smell abnormality question.
Change in Brief Smell Identification Test (B-SIT) Scores | Baseline to day 60
  The B-SIT is a shorter 12-item version of the full 40-item University of Pennsylvania Smell Identification Test (UPSIT). It is a validated 5 minute screening test for detecting smell loss. The test employs 12 well known cross cultural odors in a scratch and sniff format. Percentile norms are based upon nearly 4000 subjects via the B-SIT administration manual and both the test and the manual with a scoring key are available from Sensonics, Inc. (sensonics.com/smell-products/brief-smell-identification-test.html).

SECONDARY OUTCOMES:
Adult Eating Behavior Questionnaire (AEBQ) | Baseline, day 30, day 60
  Patient reported outcome of quality of life related to change in chemosensory function A validated, 35-item self-report measure that provides a comprehensive, convenient, and easy-to-use measure of an adult's appetite across 8 appetitive traits: Hunger (H), Food Responsiveness (FR), Emotional Over-Eating (EOE), Enjoyment of Food (EF), Satiety Responsiveness (SR), Emotional Under-eating (EUE), Food Fussiness (FF) and Slowness in Eating (SE). The AEBQ appears to be a reliable measure of appetitive traits in adults which translates well from the validated child measure (Child Eating Behaviour Questionnaire), and is unique in that it's scales assess food approach as well as food avoidance.95 Food Approach appetitive traits relevant to "Enjoyment of Food" will be assessed with 3 questions: "I enjoy eating", "I love food", and "I look forward to mealtimes". Internal reliability of the "Enjoyment of Food" subscale is 0.859 (Chronbach's alpha).
Functional Assessment of Anorexia/Cachexia Tool (FAACT) | Baseline, day 30, day 60
  Patient reported outcome of factors related to anorexia and cachexia. Functional Assessment of Anorexia/Cachexia Treatment tool contains a validated 12 question additional concerns module, in addition to the Functional Assessment of Cancer Therapy - General (FACT-G), which measures nutritional quality of life.
Euro Quality of Life (EuroQOL) | Baseline, day 30, day 60
  The EuroQOL is a self-reported generic health-related QoL (HRQoL) instrument that specifically addresses health status and has been tested among individuals with COVID-19 with taste and smell abnormality.4 It consists of five questions on mobility, self-care, usual activities, pain and discomfort and anxiety and depression with 3-point response categories (1=no problems, 2=some problems and 3=serious or extreme problems). The EQ-visual analogue scale (VAS) component of EQ-5D asks respondents to rate their overall health status from 0 (worst imaginable health) to 100 (best imaginable health).

OTHER OUTCOMES:
Daily self-monitoring | daily for 60 days
  Participants will track their taste and smell function each day as well as their use of the lactoferrin supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn J Lesser, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No